CLINICAL TRIAL: NCT02364596
Title: A Phase 1, Single-arm, Open-label Study To Confirm The Safety, Tolerability, And Immunogenicity Of A 4-antigen Staphylococcus Aureus Vaccine (sa4ag) In Healthy Adults Aged 18 To <65 Years
Brief Title: Evaluation of a Single Vaccination With a 4-Antigen Staphylococcus Aureus Vaccine (SA4Ag) in Healthy Adults Aged 18 to <65 Years
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: B3451015
Record Dates: First submitted 2015-01-08; First posted 2015-02-18 (Estimated); Last update posted 2015-04-03 (Estimated); Status verified 2015-04

CONDITIONS: Staphylococcal Infections
Keywords: Staphylococcus aureus vaccine; Staphylococcal infection
MeSH Terms: conditions — Staphylococcal Infections | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): SA4Ag vaccine
  Interventions: Biological: SA4Ag vaccine; Procedure: Blood sample

INTERVENTIONS:
Biological: SA4Ag vaccine — Subjects receive 1 intramuscular injection (0.5 mL) of the SA4Ag vaccine.
Procedure: Blood sample — Blood for immunogenicity will be collected from all subjects at various timepoints.

SUMMARY:
The purpose of this study is to evaluate the safety and immunogenicity of a single vaccination of an investigational vaccine against Staphylococcus aureus (SA4Ag) in healthy adults aged 18 to <65 years.

ELIGIBILITY:
Inclusion Criteria: 1. Evidence of a personally signed and dated informed consent document (ICD) indicating that the subject has been informed of all pertinent aspects of the study. 2. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures, including daily completion of the e-diary for 10 days after study vaccination. 3. Healthy male and female subjects, aged 18 to <65 years at enrollment, as determined by medical history, physical examination, and the clinical judgment of the investigator to be eligible for the study. Subjects with preexisting chronic medical conditions determined to be stable may be included. 4. Male and female subjects of childbearing potential and at risk for pregnancy must agree to use a highly effective method of contraception throughout the study. 5. Subject must be able to be contacted by telephone during study participation.

Exclusion Criteria: 1. Unstable chronic medical condition or disease requiring significant change in therapya or hospitalization for worsening disease within 3 months before receipt of investigational product. 2. Serious chronic medical disorders including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that in the investigator's opinion precludes the subject from participating in the study. 3. Congenital or acquired immunodeficiency disorder, rheumatologic disorder, or other illness requiring chronic treatment with known immunosuppressant medications, including monoclonal antibodies, within the year prior to enrollment or the use of systemic corticosteroids (equivalent of ≥10 mg/day of prednisone) for >14 days within 30 days prior to study enrollment. 4. History of leukemia, lymphoma, or underlying bone marrow disorder (eg, myelodysplasia, myeloma, myeloproliferative disorder) or history of bone marrow transplant. 5. Malignancy that required treatment with chemotherapy, immunotherapy, radiation therapy, or other antineoplastic target therapies within 24 months prior to study enrollment. 6. Any infection proven or suspected to be caused by S. aureus within 6 months preceding study vaccination. 7. Previous administration of S. aureus vaccine or S. aureus/Candida vaccine. 8. Any contraindication to vaccination or vaccine components, including previous anaphylactic reaction to any vaccine or vaccine-related components. 9. Bleeding diathesis or condition associated with prolonged bleeding time that would contraindicate intramuscular injection. 10. Donation of blood volume of 250 mL or greater (excluding protocol-required blood collection) or donation of plasma within 3 months prior to enrollment through conclusion of the study. 11. Receipt of blood products or immunoglobulins (including monoclonal antibodies) within 6 months before enrollment or anticipated through conclusion of the subject's participation. 12. Subjects who are investigational site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or subjects who are Pfizer employees directly involved in the conduct of the study. 13. Participation in other studies involving investigational drug(s) (Phases 1-4) within 30 days before the current study begins and/or during study participation. Participation in observational studies is permitted. 14. Pregnant female subjects; breastfeeding female subjects; male subjects with partners currently pregnant; male and female subjects of childbearing potential and at risk for pregnancy who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study. 15. Residence in a nursing home or long-term care facility or requirement for semiskilled nursing care. An ambulatory subject who is a resident of a retirement home or village is eligible for the trial. 16. Subjects with known active disease with human immunodeficiency virus (HIV), hepatitis B virus (HBV), and/or hepatitis C virus (HCV). 17. Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the subject inappropriate for entry into this study.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-01; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Number of subjects reporting local reactions (redness, swelling, and pain at the injection site) as self-reported on electronic diaries (e-diaries) for 10 days after vaccination. | 10 days
Number of subjects reporting systemic events (fever, fatigue, headache, vomiting, diarrhea, muscle pain, and joint pain) as self-reported on e-diaries for 10 days after vaccination. | 10 days
Number of subjects reporting adverse events (AEs) categorized according to the Medical Dictionary for Regulatory Activities (MedDRA). | 1 month
Number of subjects reporting serious adverse events (SAEs) categorized according to the Medical Dictionary for Regulatory Activities (MedDRA). | 1 month
Opsonophagocytic activity titers measured as geometric mean titers against S. aureus isolates | 1 month

SECONDARY OUTCOMES:
Competitive Luminex immunoassay titers summarized as geometric mean titers for S. aureus antigens | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (2):
- United States (2):
  - Broward Research Group, Hollywood, Florida
  - Miami Research Associates, South Miami, Florida

REFERENCES:
- [Derived] Begier E, Seiden DJ, Patton M, Zito E, Severs J, Cooper D, Eiden J, Gruber WC, Jansen KU, Anderson AS, Gurtman A. SA4Ag, a 4-antigen Staphylococcus aureus vaccine, rapidly induces high levels of bacteria-killing antibodies. Vaccine. 2017 Feb 22;35(8):1132-1139. doi: 10.1016/j.vaccine.2017.01.024. Epub 2017 Jan 28. PMID 28143674